CLINICAL TRIAL: NCT02123186
Title: Newborn Screening for Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201308058RIND
Record Dates: First submitted 2014-04-21; First posted 2014-04-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Newborn Screening , spinal muscular atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- newborns testing for SMA
  Interventions: Other: newborn screening test for SMA

INTERVENTIONS:
Other: newborn screening test for SMA — Routine newborn screening dried blood spots sample is used to test if missing 2 copies of SMN1 gene.

SUMMARY:
To test if the routine newborn screening dried blood spots can be used to test if missing 2 copies of SMN1 gene, a status indicating spinal muscular atrophy

DETAILED DESCRIPTION:
Parents of newborns will be invited to test if their newborns are affected with SMA. The routine newborn screening dried blood spots sample will be used to test if missing 2 copies of SMN1 gene. If positive of screening test, further confirmation tests including physical examination and other methology for SMN1 gene copies quantification will be provided. Genetic counseling and treatment option will be provided, too.

ELIGIBILITY:
Inclusion Criteria:

* Babies born in Taiwan receive regular new born screening suggested by Ministry of Heath and Welfare.
* Parents or Legal Guardian sign in the informed consent form.

Exclusion Criteria:

* Parents or Legal Guardian do not agree to sign in the informed consent form.

Ages: 2 Days to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns whose parents agree to be tested
Sampling Method: Non-Probability Sample
Enrollment: 120267 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
numbers of newborn with spinal muscular atrophy | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Hsiu Chien, M.D., PhD., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Chien YH, Chiang SC, Weng WC, Lee NC, Lin CJ, Hsieh WS, Lee WT, Jong YJ, Ko TM, Hwu WL. Presymptomatic Diagnosis of Spinal Muscular Atrophy Through Newborn Screening. J Pediatr. 2017 Nov;190:124-129.e1. doi: 10.1016/j.jpeds.2017.06.042. Epub 2017 Jul 12. PMID 28711173